CLINICAL TRIAL: NCT02633709
Title: A Single-Center, Randomized, Investigator/Subject-Blind, Adaptive Single-Ascending-Dose(SAD), Placebo-Controlled, Parallel Study to Investigate the Safety, Tolerability, Pharmacokinetics (Including the Effect of Food and the Effect of Itraconazole on the Pharmacokinetics of a Single Oral Dose of RO7034067), and Pharmacodynamics of RO7034067 Following Oral Administration in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Risdiplam (RO7034067) Given by Mouth in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP29840; 2015-004605-16 (EudraCT Number)
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Itraconazole; Risdiplam

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Part 1: Single Ascending Dose: Placebo (Placebo Comparator): Participants will receive a single dose of matching placebo orally on Day 1 of Part 1.
  Interventions: Other: Placebo
- Part 1: Single Ascending Dose: Risdiplam (Experimental): Participants will receive a single ascending dose (SAD) of Risdiplam orally on Day 1 of Part 1.
  Interventions: Drug: Risdiplam
- Part 2: Food Effect: Fasted-Fed (Experimental): This arm consists of two periods. In Period 1 participants will receive one oral dose of Risdiplam in the fasted state on Day 1. In Period 2 participants will receive one oral dose of Risdiplam in the fed state on Day 1.
  Interventions: Drug: Risdiplam
- Part 2: Food Effect: Fed-Fasted (Experimental): This arm consists of two periods. In Period 1 participants will receive one oral dose of Risdiplam in the fed state on Day 1. In Period 2 participants will receive one oral dose of Risdiplam in the fasted state on Day 1.
  Interventions: Drug: Risdiplam
- Part 3: Itraconazole Interaction (Experimental): In Period 1 a single oral dose of Risdiplam will be administered. After a wash-out period in Period 2 participants will be administered oral doses of itraconazole twice daily from Day 1 to Day 8. On Day 4 participants will receive a single oral dose of Risdiplam in the fed state in combination with itraconazole.
  Interventions: Drug: Itraconazole; Drug: Risdiplam

INTERVENTIONS:
Drug: Itraconazole — Itraconazole will be administered as an oral 200 mg dose twice daily from Day 1 to Day 8 in Part 3.
  Other Names: Sporanox®
  Arms: Part 3: Itraconazole Interaction
Other: Placebo — In Part 1 of the study matching oral placebo will be administered once on Day 1.
  Arms: Part 1: Single Ascending Dose: Placebo
Drug: Risdiplam — Single ascending oral doses of Risdiplam will be administered on Day 1 of Part 1. In Part 2 a single dose of Risdiplam will be once administered under fasted and once under fed conditions. In Part 3 a single dose of Risdiplam will be once administered alone (Period 1) and once concomitantly to itraconazole (Period 2).
  Other Names: RO7034067
  Arms: Part 1: Single Ascending Dose: Risdiplam; Part 2: Food Effect: Fasted-Fed; Part 2: Food Effect: Fed-Fasted; Part 3: Itraconazole Interaction

SUMMARY:
The objective of this study is to assess the safety and tolerability of Risdiplam (RO7034067) in healthy people. The study will assess what the body does to Risdiplam (RO7034067) and what Risdiplam (RO7034067) does to the body. Risdiplam (RO7034067) will be given by mouth in gradually increasing doses. The data from this study will help to define the dose to further explore Risdiplam (RO7034067) in patients with Spinal Muscular Atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men, aged 18 to 45 years of age, inclusive
* Body Mass Index (BMI) of 18 to 30 kilograms/meter square, inclusive

Exclusion Criteria:

* History or evidence of any medical condition potentially altering the absorption, metabolism or elimination of drugs
* History of malignancy in the past 5 years
* A history of clinically significant hypersensitivity (e.g. drugs, excipients) or allergic reactions
* Any major illness within one month before the screening examination or any febrile illness within one week prior to screening and up to first study drug administration
* History or presence of clinically significant electrocardiogram (ECG) abnormalities or cardiovascular disease
* Clinically significant abnormalities in laboratory test results
* Confirmed resting pulse rate (PR) greater than 100 or less than 40 bpm
* Confirmed systolic blood pressure (SBP) greater than 140 or less than 90 mm Hg, and diastolic blood pressure (DBP) greater than 90 or less than 50 mm Hg
* Positive result on HIV1 and HIV2, hepatitis C (HCV) or hepatitis B (HBV)
* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, ophthalmological, dermatological, hematological or allergic disease, metabolic disorder, hypofertility, cancer or cirrhosis
* History or evidence of (neuro)muscular disorders
* Hypersensitivity to itraconazole, to any of the other ingredients, or to any other triazole antifungal
* Any other known contraindications to itraconazole

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2016-08-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Parts 1 and 2: Up to 21 days after last dose of study drug. Part 3: Up to 28 days after last dose of study drug.
Percentage of Participants with Laboratory Test Abnormalities | Parts 1 and 2: Up to 21 days after last dose of study drug. Part 3: Up to 28 days after last dose of study drug.
Percentage of Participants with Clinically Significant Changes in Safety Measurements, Including Vital Signs and Electrocardiograms (ECGs) | Parts 1 and 2: Up to 21 days after last dose of study drug. Part 3: Up to 28 days after last dose of study drug.
Percentage of Participants with Clinically Significant Changes in Ophthalmological Assessments | Part 1: Up to 26 weeks; Part 2 (Treatment Period [TP] 1 and 2): Up to 29 weeks; Part 3 (TP 1, 2): Up to 30 weeks

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Time to Maximum Plasma Concentration (Tmax) | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Area Under the Plasma Concentration-Time Curve up to the Last Measurable Concentration (AUClast) | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Area Under the Plasma Concentration-Time Curve up to Time t (AUC0-t) | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Apparent Terminal Half-Life (t1/2) | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Apparent Oral Clearance (CL/F) | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Apparent Oral Volume of Distribution (Vz/F) | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Cumulative Amount Excreted Unchanged into Urine (Ae) | Part 1: Day 1, 2, 3, 4
Renal Clearance (CLR) | Part 1: Day 1, 2, 3, 4
Fraction of Dose Excreted Unchanged Renally (Fe) | Part 1: Day 1, 2, 3, 4
Metabolite-to-Parent Ratio (AUCm/AUCp) Corrected for Molecular Weight for AUCInf, AUClast or AUC0-t | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Change from In Vivo Baseline in Splicing Modifications of SMN mRNAs, Including SMN1, SMN2 FL, and SMNdelta7 mRNA in Blood Ex Vivo | Part 1: Day 1
Change from Baseline in SMN Protein Levels in Blood | Part 1: Day -1, 1, 2, 3, 4, 5, 7
Metabolite-to-Parent Ratio (Cmax_m/Cmax_p) for Cmax, Corrected for Molecular Weight | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Predose Trough Plasma Concentration (Ctrough) of Itraconazole | Parts 1 and 2: Up to Day 21; Part 3: Up to Day 28
Change from Baseline in Splicing Modifications of Survival of Motor Neuron (SMN) Messenger Ribonucleic Acids (mRNAs), Including SMN1, SMN2 FL, and SMNdelta7 mRNA in Blood In Vivo | Part 1: Day -1, 1, 2, 3, 4, 5

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Pra International Group B.V, Groningen, Netherlands

REFERENCES:
- [Derived] Cleary Y, Kletzl H, Grimsey P, Heinig K, Ogungbenro K, Silber Baumann HE, Frey N, Aarons L, Galetin A, Gertz M. Estimation of FMO3 Ontogeny by Mechanistic Population Pharmacokinetic Modelling of Risdiplam and Its Impact on Drug-Drug Interactions in Children. Clin Pharmacokinet. 2023 Jun;62(6):891-904. doi: 10.1007/s40262-023-01241-7. Epub 2023 May 6. PMID 37148485